CLINICAL TRIAL: NCT06562413
Title: Unraveling the Spectrum of Migraine Resistant to Treatments: Searching for Novel Biological PHEnotypes and theRApeutic Approaches (SPHERA Project)
Brief Title: Searching for Novel Biological Phenotypes in Migraine Patients Resistant to Treatments
Acronym: SPHERA_WP1_2
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of L'Aquila (Other)
Responsible Party: Sponsor
Other Study IDs: SPHERA-functional
Record Dates: First submitted 2024-08-08; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Migraine Disorders; Chronic Migraine; Episodic Migraine
Keywords: migraine; anti CGRP mABs; calcitonin gene related peptide; HD EEG; functional MRI; brain connectivity
MeSH Terms: conditions — Migraine Disorders | interventions — Ligands

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: Patients with high frequency episodic or chronic migraine undergoing treatment with monoclonal antibodies directed against calcitonin gene related peptide pathway (mAbs) who obtained a reduction in monthly migraine days equal or higher than 50% compared to pre-treatment values.
  Interventions: Drug: MAbs
- NON-Responders: Patients with high frequency episodic or chronic migraine undergoing mAbs treatment who obtained a reduction in monthly migraine days < 50% compared to pre-treatment values.
  Interventions: Drug: MAbs

INTERVENTIONS:
Drug: MAbs — Monthly or quarterly mAbs administration
  Other Names: Monoclonal antibody targeting the CGRP pathway (ligand or receptor) (mAbs)

SUMMARY:
The investigators aim to define the neurofunctional phenotype of migraine patients who did not respond to at least 3 preventive treatments, including monoclonal antibodies (mAbs) targeting calcitonin gene-related peptide (CGRP) pathway (NON-responders).

Primary aim will be to assess and compare changes in functional resting-state connectivity at baseline and after three months of mAbs treatment between patients who will achieve a reduction of monthly migraine days >/= than 50% (namely Responders) and those who will not (namely Responders).

The 2 groups will undergo a neurofunctional profile by means of High Density-electroencephalogram (HD-EEG) and functional-magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
High Density-electroencephalogram (HD-EEG) and functional-magnetic resonance imaging (fMRI) are widely available as powerful means to non-invasively study brain connectivity features in migraine patients.

They both enables to record brain activity with high spatial resolution. HD-EEG also contributes to high temporal resolution, while fMRI contributes to precise evaluation of deep cortical and subcortical areas, relevant in migraine pathophysiology.

Aim of the study is to evaluate changes in resting-state functional connectivity in patients undergoing preventive mAbs treatment using HD- EEG and fMRI. These findings will allow the identification of a multibiomarkers panel signature of migraine patients resisting to specifically targeted preventive treatments and potentially unveiling other molecular targets for therapeutic approaches.

STUDY DESIGN:

This study is part of the SPHERA project receiving funding from the Italian Ministry of Health (GR-2021-12372429). Patients will be enrolled from those attending the outpatient clinic of IRCCS Mondino Institute (Pavia) and Neurology Department of the University of L'Aquila (Avezzano).

The investigators will collect clinical data and perform neurofunctional profiling of migraine patients at baseline (T0) and after three months of mAbs treatment (T3).

METHODS:

All patients will undergo a resting-state functional evaluation through high density-EEG and subset of 40 patients will also be studied in parallel with fMRI at baseline.

- HD-EEG: the investigators will randomly acquire 4 recordings (6 minutes each) in resting-state condition, 2 with opened eyes, and 2 with closed eyes. The investigators will consider the following frequency bands: delta (1-4 Hz), theta (4-8 Hz), alfa (8-13 Hz), beta (13-30 Hz), gamma (30-80 Hz).

Acquisition parameters will be: High-Pass: 0.5 Hz; Low-Pass: 100 Hz; Notch: 50 Hz. For analysis of HD-EEG data, the investigators will use a tailored analysis pipe-line that was previously developed and validated to reconstruct neural sources from cortical/subcortical gray matter (Semprini, 2021). EEG signals will be band-pass filtered (1-80 Hz) and down-sampled at 250 Hz. Biological artifacts will be rejected using Independent Component Analysis (ICA). EEG signals will be referenced with a customized version of the Reference Electrode Standardization Technique (REST) (Mantini, 2007). A matrix will estimate the relationship between the measured scalp potentials and the dipoles corresponding to brain sources. Sources reconstruction will be performed with the exact low-resolution brain electromagnetic tomography (eLORETA) algorithm.

- Resting state fMRI: ICA will be applied to resting state-fMRI to characterize the RSNs. For each subject and for each identified RSN, the mean functional connectivity will be calculated. A seed based component analysis will be applied in order to obtain a whole brain map to describe the strength of the connectivity of each voxel of the brain image with the region of interest (seed). The region of interests selection will be based on available literature and previous experience.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients aged 18 to 75 years
* diagnosis of episodic migraine or chronic migraine according to ICHD-3 criteria
* for episodic migraine: 8-14 monthly migraine days in the previous 3 months
* diagnosis of resistant migraine, defined by having failed at least 3 classes of migraine preventatives and suffer from at least 8 debilitating monthly headache days for at least 3 consecutive months
* patients naive to CGRP targeting treatments

Exclusion Criteria:

* history of major psychiatric or other neurological conditions
* diagnosis of other primary or secondary headache disorders (only sporadic tension-type headache is allowed if the patients can clearly differentiate between the 2 types of headaches)
* changes in ongoing preventive treatment (if any) in the previous 3 months
* clinically significant medical conditions
* chronic pain conditions
* alcohol and/or drug abuse
* pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic and high frequency episodic migraine attending the outpatient clinic of the Headache Science & Neurorehabilitation Unit of the IRCCS Mondino Foundation (Pavia, Italy) and the Neurology Department of the University of L'Aquila (Avezzano, Italy).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
RSN-FC assessed through HD-EEG | Baseline (T0), and three months of mAbs treatment (T1)
  Resting state functional connectivity assessed through HD-EEG (continuous variable, without unit of measurement)
RSN-FC assessed through MRI | Baseline (T0)
  Resting state functional connectivity assessed through MRI (continuous variable, without unit of measurement)

SECONDARY OUTCOMES:
Comparison between baseline RSN-FC assessed through HD-EEG | Baseline (T0)
  Comparison between RSN-FC changes assessed through HD-EEG (continuous variable, without unit of measurement)
Comparison between baseline RSN-FC assessed through MRI | Baseline (T0)
  Comparison between RSN-FC changes assessed through MRI (continuous variable, without unit of measurement)

CONTACTS AND LOCATIONS:
Locations (1):
- Headache Science & Neurorehabilitation Unit, Pavia, Italy

REFERENCES:
- [Background] Mantini D, Franciotti R, Romani GL, Pizzella V. Improving MEG source localizations: an automated method for complete artifact removal based on independent component analysis. Neuroimage. 2008 Mar 1;40(1):160-73. doi: 10.1016/j.neuroimage.2007.11.022. Epub 2007 Dec 3. PMID 18155928
- [Background] Gao W, Walther A, Wekenborg M, Penz M, Kirschbaum C. Determination of endocannabinoids and N-acylethanolamines in human hair with LC-MS/MS and their relation to symptoms of depression, burnout, and anxiety. Talanta. 2020 Sep 1;217:121006. doi: 10.1016/j.talanta.2020.121006. Epub 2020 Apr 9. PMID 32498885
- [Background] Fuertig R, Ceci A, Camus SM, Bezard E, Luippold AH, Hengerer B. LC-MS/MS-based quantification of kynurenine metabolites, tryptophan, monoamines and neopterin in plasma, cerebrospinal fluid and brain. Bioanalysis. 2016 Sep;8(18):1903-17. doi: 10.4155/bio-2016-0111. Epub 2016 Aug 15. PMID 27524289
- [Background] Curto M, Lionetto L, Negro A, Capi M, Fazio F, Giamberardino MA, Simmaco M, Nicoletti F, Martelletti P. Altered kynurenine pathway metabolites in serum of chronic migraine patients. J Headache Pain. 2015;17:47. doi: 10.1186/s10194-016-0638-5. Epub 2016 Apr 29. PMID 27130315
- [Background] Greco R, Demartini C, Zanaboni AM, Tumelero E, Icco R, Sances G, Allena M, Tassorelli C. Peripheral changes of endocannabinoid system components in episodic and chronic migraine patients: A pilot study. Cephalalgia. 2021 Feb;41(2):185-196. doi: 10.1177/0333102420949201. Epub 2020 Sep 23. PMID 32967434
- [Background] De Icco R, Greco R, Demartini C, Vergobbi P, Zanaboni A, Tumelero E, Reggiani A, Realini N, Sances G, Grillo V, Allena M, Tassorelli C. Spinal nociceptive sensitization and plasma palmitoylethanolamide levels during experimentally induced migraine attacks. Pain. 2021 Sep 1;162(9):2376-2385. doi: 10.1097/j.pain.0000000000002223. PMID 33587406